CLINICAL TRIAL: NCT03262714
Title: Effects of Dancing and Walking on Cardiovascular Risk Factors and Functional Capacity in Older Women: a Randomized Controlled Trial.
Brief Title: Effects of Dancing on Cardiovascular and Functional Risk Factors in Older Women.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alvaro Reischak-Oliveira, Professor Alvaro Reischak-Oliveira, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 53834516.0.0000.5347
Record Dates: First submitted 2017-08-08; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Aging; Cardiovascular Risk Factor; Physical Activity
Keywords: Dance, walking, cardiovascular risk, functional capacity.
MeSH Terms: conditions — Motor Activity | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dancing (Experimental): Elderly women randomized to the dance intervention programme.
  Interventions: Other: Dance
- Walking (Experimental): Elderly women randomized to the walking intervention programme.
  Interventions: Other: Walking
- Stretching (Active Comparator): Elderly women randomized to the stretching intervention programme.
  Interventions: Other: Stretching

INTERVENTIONS:
Other: Dance — Participants randomized to the dance group will take part in a dance intervention programme for 8 weeks, including 3 sessions per week, each lasting 60 min. Dance classes will be performed in group in a dance studio, including a variety of rhythms such as salsa, jazz and aerobics. The dance session wil include a warm up of 15 min (posture, join mobility and dance technique), a main part of 40 min (learning of specific choreographies and practice of moves across the floor), and a cool down of 5 min (muscle stretching and relaxation).
  Arms: Dancing
Other: Walking — Participants randomized to the walking group will take part in a walking intervention programme for 8 weeks, including 3 sessions per week, each lasting 60 min. The walking session will include a warm up of 10 min (posture and join mobility), a main part of 40 min (walking on a treadmill with a heart rate corresponding to 60% of VO2peak), and a cool down of 10 min (muscle stretching and relaxation).
  Arms: Walking
Other: Stretching — Participants randomized to the control group will take part in stretching classes, once a week, each lasting 60 min, also for 8 weeks. Stretching exercises for large muscle groups will be performed standing or in a match, holding the positions for a maximum of 10 s. There will be no music playing during the session.
  Arms: Stretching

SUMMARY:
The goal of this randomized controlled trial is to investigate the effects of a dance intervention on cardiovascular risk factors and functional capacity of older women, comparing dancing to a walking exercise intervention and to an active control condition (stretching). The participants will include women between 60 and 80 years old, with body mass index inferior to 35 Kg /m2. The main outcome of this study is the peak oxygen consumption (VO2peak). The secondary outcomes are cardiovascular risk associated factors (C-reactive protein, TNF-alpha, lipid profile, etc) and functional performance (muscle strength and power, balance, gate ability, etc). The experimental design will include 3 parts: 1) Pre-intervention assessments: medical evaluation, fasting blood exams, maximum exercise test, assessments of body composition, balance, gate ability, muscular strength and power. 2) Period of interventions: patients will be randomized to one of the three following groups: dance, walking or stretching. The duration of the interventions will be 8 weeks, including 3 sessions per week for dance and walking, and once a week for the stretching group. Each session will last 60 min. 3) Post-intervention assessments: the same protocols of testing as pre-intervention.

DETAILED DESCRIPTION:
The aging process is characterized by reductions of lean mass simultaneously to increases in visceral adipose tissue. Metabolically, this is related to insulin resistance and higher risk to develop cardiovascular diseases. Functionally, loss of strength and cardiorespiratory fitness may lead to early muscle fatigue onset, which may limit the performance of daily activities, and eventually lead to loss of independence with aging. Dancing has been used as a form of exercise to improve functional and metabolic outcomes during aging. However, the field lacks of randomized controlled trials (RCT) evaluating metabolic outcomes related to dance interventions, as well as comparisons of dancing with other types of exercise on functional performance and metabolic health of older adults. Therefore, the goal of this randomized controlled trial is to investigate the effects of a dance intervention on cardiovascular risk factors and functional capacity of older women, comparing dancing to a walking exercise intervention and to an active control condition (stretching). Additionally, we aim to investigate the acute cardiorespiratory responses of a dance session. The participants will include women between 60 and 80 years old, with body mass index inferior to 35 Kg /m2 and independent for performing daily activities. They should not be engaged in any type of regular physical activity in the past 6 months. Exclusion criteria will include type 2 diabetes mellitus, cardiovascular complications and neurodegenerative diseases. The main outcome of this study is the peak oxygen consumption (VO2peak), as it has been associated with both, cardiovascular risk and functional performance in aging individuals. The secondary outcomes are: (1) cardiovascular risk associated factors: C-reactive protein, TNF-alpha, triglycerides, total cholesterol, LDL-cholesterol, HDL-cholesterol, fasting glucose and insulin, and homeostatic model assessment of insulin resistance (HOMA-IR). (2) Functional performance: muscle strength and power, balance, gate ability and muscle quality. The experimental design will include 3 parts: 1) Pre-intervention assessments: medical evaluation, fasting blood exams, maximum exercise test, assessments of body composition, balance, gate ability, muscular strength and power. 2) Period of interventions: patients will be randomized in blocks (randomization.com), in accordance to their VO2peak , to one of the three following groups: dance, walking or control. The duration of the dance and walking interventions will be 8 weeks, including 3 sessions per week, each lasting 60 min. Dance classes will be performed in group in a dance studio, including a variety of rhythms such as salsa, jazz and aerobics. Walking sessions will be performed individually or in groups of two people, in a treadmill, at the gym. The control group will have 60min stretching classes once a week, also for 8 weeks. 3) Post-intervention assessments: the same protocols of testing of the pre-interventions assessments will be repeated. All the assessments and interventions will be held at the Laboratory of Research in Exercise (LAPEX-UFRGS).

ELIGIBILITY:
Inclusion Criteria:

* Women between 60 and 80 years old
* BMI inferior to 35 kg/m2
* Independent for performing daily activities (OARS scale)
* Not engaged in any type of regular exercise programme for the past 6 months

Exclusion Criteria:

* Type 2 diabetes mellitus, dyslipidemia, cardiovascular diseases or other non-controlled metabolic disorders
* Chronic diseases such as fibromyalgia, cancer or neurodegenerative disorders
* Bone, joints or muscle problems that could impair exercise performance
* Not being able to perform the effort test in the first assessment session, abnormal electrocardiogram, or any other condition identified by the physician of the study that limit the engagement in an exercise training programme.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Oxygen Consumption (VO2peak) | Baseline and 8 weeks
  The maximum capacity of oxygen consumption measured during an incremental exercise test.

SECONDARY OUTCOMES:
Change in C-reactive protein (CRP) | Baseline and 8 weeks
  Cardiovascular risk marker. It will be analyzed in plasma, using ELISA specific kits.
Change in Tumor necrosis factor alpha (TNF-alpha) | Baseline and 8 weeks
  Inflammatory marker. It will be analyzed in plasma, using ELISA specific kits.
Change in Triglycerides | Baseline and 8 weeks
  Lipid profile marker. It will be analyzed in plasma, by enzymatic colorimetric method, using an automatic analyzer (ROCHE, Cobas C111, Switzerland).
Change in Total Cholesterol | Baseline and 8 weeks
  Lipid profile marker. It will be analyzed in plasma, by enzymatic colorimetric method, using an automatic analyzer (ROCHE, Cobas C111, Switzerland).
Change in LDL-Cholesterol | Baseline and 8 weeks
  Lipid profile marker. Estimation of the LDL concentration will be calculate using the formula of Friedewald.
Change in HDL-Cholesterol | Baseline and 8 weeks
  Lipid profile marker. It will be analyzed in plasma, by enzymatic colorimetric method, using an automatic analyzer (ROCHE, Cobas C111, Switzerland).
Change in Fasting Glycemia | Baseline and 8 weeks
  Glycaemic profile marker. It will be analyzed in plasma, by enzymatic colorimetric method, using an automatic analyzer (ROCHE, Cobas C111, Switzerland).
Change in Fasting Insulin | Baseline and 8 weeks
  Glycaemic profile marker. It will be measured in plasma, usin a high sensitivity enzyme-linked immunosorbent assay.
Change in HOMA-IR | Baseline and 8 weeks
  Glycaemic profile marker. Homeostatic model of insulin resistance. It will be calculated according to the following formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
Change in Muscle Strength | Baseline and 8 weeks
  Isometric peak torque of the knee extensors will be measured using an isokinetic dynamometer (Cybex Norm, EUA).
Change in Muscle Power | Baseline and 8 weeks
  Lower body muscle power will be measured by the performance of the counter movement jump in a force platform.
Change in Muscle Quality | Baseline and 8 weeks
  Echo intensity of the quadriceps will be analyzed by ultrasound images.
Change in Static Balance | Baseline and 8 weeks
  Static balance will be measured by a single leg support balance test, performed with both legs, with the eyes open and closed.
Change in Dynamic Balance | Baseline and 8 weeks
  Dynamic balance will be measured by the Time to Up ang Go (TUG) test.
Change in Gate ability | Baseline and 8 weeks
  Gate ability will be measured in a 10m track, picking up objects and passing over obstacles.
Change in Body Weight | Baseline and 8 weeks
  Measurements of body weight will be measured in a digital scale.
Change in Waist Circumference | Baseline and 8 weeks
  Measurements of waist circumference will be performed with a measuring tape.
Change in Percentage of Body Fat | Baseline and 8 weeks
  Measurements of skinfolds will be taken to calculate the percentage of body fat.
Change in Sit and Stand ability | Baseline and 8 weeks
  The ability to sit and stand in a chair 5 times, as fast as possible.
Changes in Fall Risk | Baseline and 8 weeks
  The risk of fall will be measured by the performance in the TUG test.
Changes in the Fear of Falling | Baseline and 8 weeks
  The fear of falling will be analyzed by the Falls Efficacy Scale-International Brazil (FES-I-Brazil).
Changes in Quality of Life | Baseline and 8 weeks
  Quality of life will be analyzed by the questionary WHOQOL (World Health Organization Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Reischak-Oliveira, PhD., Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Rodrigues-Krause J, Farinha JB, Ramis TR, Macedo RCO, Boeno FP, Dos Santos GC, Vargas J Jr, Lopez P, Grazioli R, Costa RR, Pinto RS, Krause M, Reischak-Oliveira A. Effects of dancing compared to walking on cardiovascular risk and functional capacity of older women: A randomized controlled trial. Exp Gerontol. 2018 Dec;114:67-77. doi: 10.1016/j.exger.2018.10.015. Epub 2018 Oct 31. PMID 30389581